CLINICAL TRIAL: NCT02644629
Title: Intra-nasal vs. Intra-venous Ketamine Administration as an add-on to Antidepressant Therapy
Brief Title: Intra-nasal vs. Intra-venous Ketamine Administration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Principal Investigator, Aviv Segev, Head, Psychiatric Emergency Services, Shalvata Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHA-15-0019
Record Dates: First submitted 2015-12-27; First posted 2016-01-01 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sodium Chloride; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active IV (Active Comparator): Will receive IV Ketamine, along with IN placebo.
  Interventions: Drug: Placebo; Drug: Ketamine (1st phase); Drug: Ketamine (2st phase)
- Active IN (Active Comparator): Will receive IN Ketamine, along with IV placebo.
  Interventions: Drug: Placebo; Drug: Ketamine (1st phase); Drug: Ketamine (2st phase)

INTERVENTIONS:
Drug: Placebo — Saline 0.9%, Administration of 0.2mg/kg (IV Push) or 50mg (IN, 5 doses, alternating nostrils)
  Other Names: Saline 0.9%
Drug: Ketamine (1st phase) — Administration of 0.2mg/kg (IV Push) or 50mg (IN, 5 doses, alternating nostrils)
  Other Names: Ketalar
Drug: Ketamine (2st phase) — Patients failing to achieve response (<50% MADRS score) in the parallal phase, will be offered additional 4 session (twice a week, 2 weeks) of 0.5 mg/kg ketamine over 40 minutes.
  Other Names: Ketalar

SUMMARY:
The current study wishes to contribute to the applicability of the use of ketamine in a clinical setting by focusing on the efficacy of intra-nasal administration compared with the IV route.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Diagnosis of MDD (Major Depressive Disorder), made or affirmed by a senior psychiatrist in Shalvata
3. MADRS score > 20
4. Treated with conventional anti-depressant, administered within a formal psychiatric clinic or by a certified psychiatrist.

Exclusion Criteria:

1. Active or past psychotic disorder, including a history of psychotic affective state
2. Mental Retardation or Autistic Spectrum Disorder
3. Prominent personality disorder
4. Cardiac or neurologic active medical condition, including past CVA/TIA (Cardiovascular Accident/Transient Ischemic Attack) or any other unstable medical condition.
5. Chronic nasal congestion
6. Active or recent drug or alcohol abuse
7. Substantial suicidality in a patient requiring admission but refuses to do so, and signs an "against medical advice" release form as part of clinical evaluation, and does not answer the terms for involuntary admission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
MADRS (Montgomery-Åsberg Depression Rating Scale) score improvement from baseline | 15 weeks

SECONDARY OUTCOMES:
Ratio of subjects achieving remission | 15 weeks
Ratio of subjects achieving Response | 15 weeks
Durability of anti-depressant effect according to MADRS Score | 15 weeks
  The rate of effect decline, as measured by MADRS Questionnaire
Tolerability of Route, based on side effects questionnaire | 3 weeks
  Adverse side effects reported by subjects, as reported in side effects questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aviv Segev, MD, Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel